CLINICAL TRIAL: NCT00512629
Title: Cholestasis Prevention: Efficacy of IV Fish Oil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Puder, Medical Staff, Boston Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-03-0105; 1R01FD003436-01 (FDA)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Cholestasis; Parenteral Nutrition
Keywords: PN; cholestasis; gastrointestinal disease in infants; short bowel syndrome
MeSH Terms: conditions — Cholestasis; Hyperphagia; Short Bowel Syndrome | interventions — fish oil triglycerides; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omegaven (Experimental): Omegaven is a fish based intravenous fat emulsion
  Interventions: Drug: Omegaven
- Intralipid (Active Comparator)
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: Omegaven — Omegaven is a fish based intravenous fat emulsion
  Arms: Omegaven
Drug: Intralipid — Intralipid is a plant based intravenous fat emulsion
  Arms: Intralipid

SUMMARY:
Parenteral nutrition (PN) solutions are life saving in patients with surgical gastrointestinal diseases. However, the use of PN in pediatric populations, especially premature infants, is frequently associated with liver injury that may ultimately result in hepatic failure. In studies conducted in a murine model, we observed that intravenous fat emulsions (IFE) comprised of omega-3 fatty acids were able to prevent the development of cholestasis, a common precursor of PN-associated liver disease, as well as reverse preexisting PNALD through a combination of factors, including improved triglyceride clearance coupled with anti-inflammatory properties. In a case series treating patients with hepatic cholestasis, serum bilirubin levels decreased markedly after the parenteral administration of an omega-3 fatty acid based fat emulsion (Omegaven®). Patients tolerated this therapy and no adverse reactions attributed to its use were observed. Based on results of these previous studies, we propose to conduct a randomized trial aiming to gain preliminary evidence of efficacy of an omega-3 fatty acid based IFE in preventing PNALD in children with intestinal failure

DETAILED DESCRIPTION:
We propose to conduct a randomized controlled clinical trial to determine whether the use of an omega-3 fatty acid based IFE in infants with surgical gastrointestinal disease will improve clinical outcomes compared to infants treated with standard IFE up to 6 months post randomization. Neonates and infants < 3 months old (postnatally) with surgical gastrointestinal disease (defined as congenital or acquired gastrointestinal disease requiring PN for more than 21 days) will be eligible for enrollment. Patients who meet all inclusion and exclusion criteria will be randomized to receive PN with either Intralipid® or Omegaven®. The appearance of both IFEs is indistinguishable, so patients, families and the medical care team will be blinded to treatment group allocation. Aside from the IFE type, the clinical care of both groups of infants will remain unchanged, including standard use of feeding advancement protocols, and treatment of underlying gastrointestinal and other diseases.

ELIGIBILITY:
Inclusion criteria (all of the following):

1. Congenital or acquired gastrointestinal disease requiring surgical intervention [such as Midgut volvulus, Gastroschisis-(with known or suspected atresia(s), perforation(s) requiring a jejunostomy, or bowel resections > 20cm), Omphalocele, Jejunal atresia or NEC-(no peritoneal drains) or duodenal atresia] ; and
2. Expected dependence on parenteral nutrition for full or partial nutritional support for an anticipated duration of therapy of at least 21 days; Subjects will be judged by their clinical team to require PN support a minimum of 21 days based on the following criteria: inability to tolerate enteral feedings, lack of audible bowel sounds, contraindications to initiation of enteral feedings (e.g., grossly bloody stools or other sign of intestinal ischemia, hypotension, bilious emesis, or clinical or radiographic evidence of bowel obstruction); and
3. Neonates and infants < 3 months of age (postnatally); and
4. Gestational age > 28 weeks; and
5. Baseline direct bilirubin less than 1.0 mg/dL (normal); and
6. Weight > 1 kg

Exclusion criteria(any one of the following):

1. Exposure to soybean oil fat emulsion for greater than three weeks (>21 days) at time of enrollment
2. Known or suspected intolerance or allergy to any of the components of the study IFE, including fish, soy or egg protein
3. Inability to obtain written informed consent prior to the baseline labs
4. The patient is enrolled in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
5. Intention to transfer care to another patient facility within 3 months of baseline labs
6. Any serum triglyceride level greater than 400 mg/dL at baseline
7. History of severe hemolytic disorders or INR greater than 1.5 at baseline (INR cutoff of greater than 2 for babies less than 1 week of age)
8. History of shock requiring vasopressors (dopamine equal or less than 20 micrograms/kilogram/minute is allowed; all other use of vasopressors is excluded)
9. Preexisting liver disease, regardless of etiology
10. Hemodynamically unstable as judged by PI
11. Renal failure (creatinine greater than 0.4 mg/dL unless less than 1 month of age-then at the PI's discretion)
12. Patient previously had STEP (Serial Transverse Enteroplasty Procedure)
13. Patient is currently on ECMO or nitric oxide
14. GGTP > 80 mg/L at baseline
15. Weight < 1 kg at time of enrollment
16. Gestational age < 28 weeks at time of enrollment

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Presence vs. absence of PN-associated cholestasis (PNAC) | 6 months
  The definition of "Presence vs. Absence of PNAC" will vary with the post conceptual age of the child. In infants > 40 weeks post conceptual age, we will define PN-associated cholestasis as four consecutive measurements (> 6 days apart) of serum direct bilirubin > 2.0mg/dL obtained over a 30 day period in the absence of other demonstrable etiologies of cholestasis. Due to hepatic immaturity, for infants < 40 weeks post conceptual age, PN associated cholestasis will be defined as four consecutive measurements (> 6 days apart) of serum direct bilirubin > 2.0mg/dL obtained over a 42 day period.

SECONDARY OUTCOMES:
Fatty acid profiles | 6 months
  (i.e., Mead acid levels, triene:tetraene ratios, total omega-3 and omega-6 fatty acid levels, arachidonic acid levels)
Weight and height gain | 6 months
Liver function tests | 6 months
  (i.e. serum triglycerides, cholesterol, ALT, AST and total and direct bilirubin levels)
Death from PNALD liver or liver/gastrointestinal tract transplant. | 1 year
Duration of parenteral nutrition | 6 months
  (i.e. enteral feeding tolerance, including days to reach full enteral feeding (approximately 100-125kcal/kg/d + 10%) after randomization and the number of episodes of feeding intolerance (defined as an interruption of enteral feedings for > 12 hrs) , number of infants requiring TPN providing > 10% of total daily fluid volume at 12 weeks after randomization, and duration of TPN providing > 10% of total daily fluid intake)
Frequency of blood stream infections | 6 months
Inflammatory markers (C-reactive protein), cytokine levels | 6 months
Incidence and severity of ROP | 6 months
Neurodevelopment Assessments | 6, 12, & 24 months (corrected for gestational age)
  Neurodevelopment will be assessed at 6, 12, and 24 months (corrected) using Bayley Scales of Infant Development III(mean total, cognitive, language, and motor scaled score; and frequency of each score <70). The MSD parent questionnaire will be mailed at 12 and 24 months (corrected); and the Parent Report of Children's Abilities - Revised (PARCA-R) parent questionnaire will be mailed at 24 months (coorected).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Puder, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Childrens's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Nehra D, Fallon EM, Potemkin AK, Voss SD, Mitchell PD, Valim C, Belfort MB, Bellinger DC, Duggan C, Gura KM, Puder M. A comparison of 2 intravenous lipid emulsions: interim analysis of a randomized controlled trial. JPEN J Parenter Enteral Nutr. 2014 Aug;38(6):693-701. doi: 10.1177/0148607113492549. Epub 2013 Jun 14. PMID 23770843